CLINICAL TRIAL: NCT02721472
Title: Plasma DNA and Vascular Remodelling in Patients With Sickle Cell Disease
Acronym: PADRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Theravia (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DRE-FR-15-1
Record Dates: First submitted 2016-03-18; First posted 2016-03-29 (Estimated); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- sickle cell disease patients (Other): Sickle cell disease patients included in the study and Plasma DNA levels will be analyzed and compared in patients with a reactive hyperaemia index (RHI) < 1.67 (endothelial dysfunction) assessed by Endo-PAT 2000 versus those recorded in patients with a RHI ≥ 1.67 (no endothelial dysfunction).
  Interventions: Procedure: micro- and macro-circulatory vascular remodelling measures not practice in routine care; Procedure: Biological measures not practice in routine care

INTERVENTIONS:
Procedure: micro- and macro-circulatory vascular remodelling measures not practice in routine care — Vascular measures : reactive hyperaemia index (RHI) assessed by Endo-PAT, central aortic blood pressure, aortic augmentation index, carotid-femoral pulse wave velocity
Procedure: Biological measures not practice in routine care — Biological measures : Plasma DNA level, NETs (plasma nucleosome levels), Microparticules (MPs) (total, associated with red blood cells, neutrophils, platelets), haem (total and bound to MPs), Myeloperoxydase and elastase activity, neutrophils/DNA, Annexin A5, RNA and TSP1

SUMMARY:
The purpose of this study is to evaluate the relationship between plasma DNA levels and micro- and macro-circulatory vascular remodelling in patients with sickle cell disease

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Homozygous SS or Sß0 sickle cell disease patients.
* Seen in consultation for an annual clinical and para-clinical evaluation of his/her disease.
* Stable clinical condition of the disease defined as the absence of severe vaso-occlusive crises (requiring hospitalisation or a visit to the emergency unit) in the previous month and absence of transfusion in the previous 3 months.

Exclusion Criteria:

* Other haemoglobinopathy
* Known diabetes.
* Recent administration of an anticoagulant treatment at curative doses (< 48h before inclusion), or platelet-inhibiting drugs (less than 1 week prior to inclusion).
* Recent transfusion (less than 3 months prior to inclusion).
* Pregnancy or post-partum (first 40 days after giving birth).
* Recent consumption of alcohol (less than 10h), coffee (less than 3h), and tobacco (less than 36h) before inclusion.
* Known infection with hepatitis B, C, and HIV infection.
* Known cancer or progressive blood disease.
* Known haemostasis or coagulation disorders.
* Progressive inflammatory or infectious diseases.
* Recent history (dating less than 3 months) of venous (pulmonary embolism, deep venous thrombosis) or arterial (acute coronary syndrome, stroke, peripheral arterial ischaemia) thromboembolic event.
* Adult patients subject to legal protection measures.
* Patients already involved in a therapeutic protocol.
* Patients not affiliated to a social security system.
* Non-inclusion criteria related to the technical requirements of the Endo-PAT:

  * Known cardiac arrhythmia.
  * Severe Raynaud's syndrome.
  * Hand or arm deformity that prevents an EndoPAT analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-05-17 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2019-11-14 (Actual)

PRIMARY OUTCOMES:
Comparison of plasma DNA levels in patients with a reactive hyperaemia index (RHI) < 1.67 (endothelial dysfunction) assessed by Endo-PAT 2000 versus those recorded in patients with a RHI ≥ 1.67 (no endothelial dysfunction) | 1 days

SECONDARY OUTCOMES:
Relationship between plasma DNA levels and cerebral micro- and macro-angiopathy assessed by CT angiography or MRI angiography and transcranial Doppler ultrasound | 1 day
Relationship between plasma DNA levels and cardiac damages | 1 day
Relationship between plasma DNA levels and pulmonary blood pressure | 1 day
Relationship between plasma DNA levels and macrocirculatory vascular measurements | 2 days
Relationship between plasma DNA levels and nephropathy | 1 day
Relationship between plasma DNA levels and a clinical index of the sickle cell disease severity in a stable condition | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: LE JEUNE Sylvain, MD, Principal Investigator — Hôpital Avicenne
Locations (1):
- Hôpital Avicenne, Bobigny, Île-de-France Region, France